CLINICAL TRIAL: NCT06250556
Title: Creatine Supplementation in Young and Elite Female Football Players
Brief Title: Creatine Supplementation for Female Football
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: creatineforwomen
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Athletes
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: pre-to-post design for experiment 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- creatine supplementation (Experimental)
  Interventions: Dietary Supplement: creatine

INTERVENTIONS:
Dietary Supplement: creatine — creatine supplementation (Creapure)

SUMMARY:
Creatine is an effective, inexpensive, and safe dietary supplement, which has been largely used in sports and clinical populations. However, creatine is much less studied in female athletes, with long-term data being particularly scant. This study aims to expand our knowledge on the effects of creatine supplementation in young (Under-20) and elite female football players. This study will comprise two experiments. The first one will be a randomized, controlled trial in which young athletes will be assigned into either creatine or placebo (n = 20). Before and 7 days after supplementation or placebo (4 x 5 g/d of Creapure or dextrose at same dose), athletes will perform a battery of performance tests. Blood and urinary biochemical parameters for assessing the safety of supplementation will be analyzed (creatinine, albuminuria, urea, sodium, potassium, liver enzymes, creatine kinase, hematology). Food intake will be assessed by means of 3-d 24-h dietary recalls. The second experiment will have a quasi-experimental design (i.e., pre-to-post), in which both young and elite football players (n = 70) will be supplemented with creatine (4 x 5 g/d for 7 days and then 5 days during the follow-up) and will be assessed for safety using the above-mentioned markers during the regular football season (~12 months). Assessments will be carried out at baseline, in the mid-season and after the season.

ELIGIBILITY:
Inclusion Criteria:

* female football players

Exclusion Criteria:

* age under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
kidney function | baseline and after the sport season (~12 months)
  serum creatinine levels

SECONDARY OUTCOMES:
kidney function | baseline and after the sport season (~12 months)
  urinary creatinine levels
kidney function | baseline and after the sport season (~12 months)
  serum urea levels
kidney function | baseline and after the sport season (~12 months)
  serum sodium levels
kidney function | baseline and after the sport season (~12 months)
  serum potassium levels
muscle damage | baseline and after the sport season (~12 months)
  serum creatine kinase levels
hemogram | baseline and after the sport season (~12 months)
  platelet count
hemogram | baseline and after the sport season (~12 months)
  red blood cell count
hemogram | baseline and after the sport season (~12 months)
  white blood cell count
hemogram | baseline and after the sport season (~12 months)
  erythrocyte sedimentation rate

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - School of Medicine of the University of Sao Paulo, São Paulo, Sao Paulo / SP
  - School of Medicine, University of Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code